CLINICAL TRIAL: NCT00961324
Title: A Randomised, Single-centre, Double-blind, Parallelgroup, Multiple Dose Trial Comparing the Within-subject Variability of SIBA and Insulin Glargine With Respect to Pharmacodynamic Response at Steady State Conditions in Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating the Within-subject Variability of NN1250 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1991; 2008-008308-42 (EudraCT Number)
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IGlar (Experimental)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — The dose level will be 0.4 units per kg body weight injected subcutaneously (under the skin) once daily for 12 days
  Arms: IDeg
Drug: insulin glargine — The dose level will be 0.4 units per kg body weight injected subcutaneously (under the skin) once daily for 12 days
  Arms: IGlar

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to evaluate the variability in the blood glucose-lowering effect of NN1250 (insulin degludec) in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 years (both inclusive)
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-07-27 (Actual); Primary Completion 2009-10-26 (Actual); Study Completion 2009-10-26 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval at steady state | 0-24 hours (derived on treatment days 6, 9 and 12)

SECONDARY OUTCOMES:
Area under the NN1250 concentration-time curve during one dosing interval at steady state | 0-24 hours (derived on treatment days 6, 9 and 12)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Hermanski L, Nosek L, Feldman A, Rasmussen S, Haahr H. Insulin degludec: four times lower pharmacodynamic variability than insulin glargine under steady-state conditions in type 1 diabetes. Diabetes Obes Metab. 2012 Sep;14(9):859-64. doi: 10.1111/j.1463-1326.2012.01627.x. Epub 2012 Jun 7. PMID 22594461
- [Result] Heise T, Korsatko S, Nosek L, Coester HV, Deller S, Roepstorff C, Segel S, Kapur R, Haahr H, Hompesch M. Steady state is reached within 2-3 days of once-daily administration of degludec, a basal insulin with an ultralong duration of action. J Diabetes. 2016 Jan;8(1):132-8. doi: 10.1111/1753-0407.12266. Epub 2015 Mar 24. PMID 25581159
- [Result] Heise T, Kaplan K, Haahr HL. Day-to-Day and Within-Day Variability in Glucose-Lowering Effect Between Insulin Degludec and Insulin Glargine (100 U/mL and 300 U/mL): A Comparison Across Studies. J Diabetes Sci Technol. 2018 Mar;12(2):356-363. doi: 10.1177/1932296817731422. Epub 2017 Sep 26. PMID 28946756
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com